CLINICAL TRIAL: NCT07212361
Title: Infant Microbiota Restoration With Maternal Microbes
Acronym: MaMi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Katri Korpela, Associate Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HUS/617/2025/71
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-08

CONDITIONS: Infant, Newborn; Gut -Microbiota; Gut Dysbiosis; Cesarean Delivery Affecting Newborn; Cesarean Section; Vaginal Delivery; Gastrointestinal Microbiota; Microbiota, Cesarean Section, Probiotics, Dysbiosis; Feces; Delivery, Obstetric; Microbiota; Microbiology; Humans; Pregnancy; Neonate
Keywords: Infant; newborn; cesarean section; neonate; restore; gut microbiota
MeSH Terms: conditions — Dysbiosis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Probiotic (Active Comparator): The infants will receive a mixture of probiotic strains currently on the market and with known safety profiles and beneficial effects on infant gut microbiota.
  Interventions: Dietary Supplement: Probiotic
- Vaginal delivery (No Intervention)
- Maternal bacteria set 1 (Experimental): The infants will receive a micture of bacteria isolated from a fecal sample of the infants' own mother.
  Interventions: Dietary Supplement: Probiotic
- Maternal bacteria set 2 (Experimental): The infants will receive a mixture of bacterial species with increased diversity isolated from the mother's sample.
  Interventions: Dietary Supplement: Probiotic
- Maternal bacteria set 3 (Other): The infants will receive a mixture of bacterial strains isolated from other infants' and/or mothers' samples to test whether bacteria from an unrelated donor have different effects compared to maternal bacteria. In this group all infants will receive the same standardised mixture of bacterial strains.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): C-section born infants given a placebo treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Specific infant-adapted commercially available strains or strains isolated from the infant's mother.
  Arms: Maternal bacteria set 1; Maternal bacteria set 2; Maternal bacteria set 3; Probiotic
Other: Placebo — Infant formula without bacteria.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test the ability of different bacterial products in restoring natural gut microbiota in C-section born infants. The main question it aims to answer is:

Do maternally derived strains of bacteria perform better than commercially available probiotic strains in restoring the gut microbiota of C-section born infants? Researchers will compare the gut microbiota of treated infants to that of untreated C-section born infants and untreated vaginally born infants to see if the bacterial treatments cause the microbiota to resemble that of vaginally born infants.

Participants will be given a bacterial product orally once daily for either one or four weeks and be asked to collect faecal, urine and saliva samples.

DETAILED DESCRIPTION:
The gut microbiota has long-term effects on host health especially in early life. Infants receive maternal faecal microbes during vaginal birth, which is prevented by C-section. C-section is associated with increased risk of many chronic diseases, likely because of the disturbed gut microbiota. We recently showed the effectiveness of a faecal microbiota transplant from the infant's own mother in restoring normal gut microbiota in C-section born infants. However, FMT contains a large diversity of unknown microbes, some of which may pose a risk of dangerous infection. A safe and widely applicable infant microbiota restoration method is urgently needed. In this project, we develop a selective microbiota transplant from mother to infant and test its efficacy and safety in a clinical trial. The work is conducted in the Faculty of Medicine, University of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mother and healthy pregnancy
* Singleton pregnancy,
* Mothers who speak Finnish or Swedish
* Mothers who are planning to breastfeed or give breastmilk by bottle to the infant
* Infants who are expected to be healthy and who will not require BCG vaccination.

Exclusion Criteria:

* Participants who lives further than a 2-hour drive from Meilahti, Helsinki, Finland
* Mothers who are not planning to breastfeed or feed breastmilk by bottle to the infant
* Mothers who are diagnosed with gestational diabetes, pre-eclampsia or who have been receiving antibiotics during the pregnancy or delivery
* Premature infants born before the pregnancy week 37
* Infants, who are born by urgent cesarean section or emergency cesarean section
* Infants, who receive antibiotics during the first week of life
* Infants, who are diagnosed with a disease, congenital anomaly or who receive less than 9 Apgar points at 5 minutes.
* Infants, who receive BCG-vaccine

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota composition, relative and absolute abundances | 1 week, 5 weeks, 11 weeks, 26 weeks and 52 weeks.
  Similarity of the overall gut, mouth, and skin microbiota composition
Fecal metabolite profiles | 1 week, 5 weeks, 11 weeks, 26 weeks and 52 weeks
  Fecal metabolite profiles in the treatment groups compared to the vaginally born reference group.

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - University of Helsinki, Helsinki

IPD SHARING:
Plan to Share IPD: No